CLINICAL TRIAL: NCT04409444
Title: An Observational Cohort Study Investigating the Impact of Community-based Lung Cancer Screening Across a Deprived Geographical Area and the Role of Biomarkers for the Early Detection of Lung Cancer.
Brief Title: Manchester Lung Health Study
Acronym: qUEST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Cancer Research UK (Other); University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: B00212; 252263 (IRAS) (Other: Health Research Authority); 19/LO/0404 (REC) (Other: Health Research Authority)
Record Dates: First submitted 2020-05-21; First posted 2020-06-01 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Environmental Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample of up to 50mL will be taken from participants for analysis of circulating tumour cells, circulating nucleic acid, proteins and genetic variations (single nucleotide polymorphisms).
  Nasal swab and brush samples will be taken for the identification of inflammatory markers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Data (main study): This study group is for any individual that attends and has a lung health check. The data collected for this study group is to evaluate the uptake and performance of a community-based lung health check / lung screening programme.
  Interventions: Diagnostic Test: Lung Cancer Screening
- Biomarker (sub-study): This sub-study is for participants that are determined to require a CT scan through their lung health check and have also signed up to the data part of the study. This part of the study is to evaluate the potential for biomarkers to improve the early detection of lung cancer.
  Interventions: Diagnostic Test: Lung Cancer Screening; Diagnostic Test: Biomarkers

INTERVENTIONS:
Diagnostic Test: Lung Cancer Screening — The lung health check consists of a symptom questionnaire for the calculation of 6-year lung cancer risk (using the PLCOM2012 model)
Diagnostic Test: Biomarkers — This will explore the role of biomarkers for the early detection of lung cancer. These include circulating nucleic acids, circulating proteins, circulating tumour cells and inflammatory markers.
  Groups: Biomarker (sub-study)

SUMMARY:
The Manchester Lung Health Study (qUEST) will assess the uptake of a community-based lung cancer screening service and its impact across a deprived area of North and East Manchester, which has high rates of lung cancer. One measure will be to compare the number and stage of lung cancers detected through screening to those detected outside of screening. In addition we will investigate the potential of a blood and nose test to detect lung cancer or to help decide who would benefit from screening. We will also see if these samples can help with the interpretation of CT scans. One of the problems with lung cancer CT screening is that you detect lung nodules in which we are not sure if they are benign or cancerous. Therefore we are also looking to see if a biomarker can help us work out which are cancerous and which are benign.

ELIGIBILITY:
Main data study:

Inclusion Criteria:

- Any individual attending the Manchester Lung Health service who has a lung health check as they meet the service inclusion exclusion criteria (see below):

Manchester Lung Health service inclusion criteria:

* Age 55-80
* Ever smoker
* Registered with a GP in the North or East Manchester area

Manchester Lung Health service exclusion Criteria:

* Lung cancer diagnosis within 5 years
* Listed on a palliative care register
* Chest CT scan within 3 months

Exclusion Criteria:

- Unable to give informed consent to study participation.

Biomarker sub-study:

Inclusion Criteria:

* Any individual attending the M-LHC service who is eligible and agrees to undergo LDCT screening.
* Has consented to the main study.

Exclusion Criteria:

* Unable to give informed consent to study participation
* Decline participation in LDCT lung cancer screening
* Known blood borne virus e.g. HIV or Hepatitis B, C

Ages: 55 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals will be attending a lung health check as they are registered to a GP practice in north and east Manchester, between the ages of 55-80 and an ever smoker.
Sampling Method: Non-Probability Sample
Enrollment: 9730 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of the Manchester lung health check service | Over 3 years to determine long term outcomes from screening
  The overall uptake will be assessed and analysed according to age, sex, smoking status, ethnicity and socio economic status.
Evaluation of biomarkers | Over 3 years to determine long term outcomes from screening
  Sensitivity and specificity of a biomarker or panel of biomarkers to detect early stage lung cancer.

SECONDARY OUTCOMES:
Screening adherence | Over 3 years to determine long term outcomes from screening
  overall and according to patient characteristics (age, sex, smoking status, ethnicity and socio economic status).
Evaluation of screening numbers required to detect lung cancer | Over 3 years to determine long term outcomes from screening
  Number needed to screen to detect one lung cancer according to lung cancer risk (as calculated by PLCOM2012).
Comparison between cohort and those residents diagnosed in north and east manchester | Over 3 years to determine long term outcomes from screening
  Lung cancer stage in the screened cohort compared to lung cancers diagnosed in residents of N+EM outside of the screening service.
Histological subtype for lung cancer related to screening service | Over 3 years to determine long term outcomes from screening
  Histological subtype of lung cancers in screening and outside of screening during the course of the service.
Treatment for lung cancer related to screening service | Over 3 years to determine long term outcomes from screening
  Treatment of lung cancers in screening and outside of screening during the course of the service.
Diagnosis route for lung cancer related to screening service | Over 3 years to determine long term outcomes from screening
  Route to diagnosis of lung cancers in screening and outside of screening during the course of the service.
False positive rates | Over 3 years to determine long term outcomes from screening
  False positive rates in those undergoing LDCT screening.
False negative rates | Over 3 years to determine long term outcomes from screening
  False negative rates in those undergoing LDCT screening.
Rates of investigation of benign disease | Over 3 years to determine long term outcomes from screening
  Rates of investigation of benign disease in those undergoing LDCT screening.
Benign resection rate in participants | Over 3 years to determine long term outcomes from screening
  Benign resection rate in participants for those that have undergoing LDCT screening.
Interval cancers | Over 3 years to determine long term outcomes from screening
  Interval cancers in those undergoing LDCT screening.
Recall rates | Over 3 years to determine long term outcomes from screening
  Recall rates in those undergoing LDCT screening.
Resection rates generated from screening | Over 3 years to determine long term outcomes from screening
  Resection rates generated from screening including incidental findings.
Investigations generated from screening | Over 3 years to determine long term outcomes from screening
  Investigations generated from screening including incidental findings.
Adverse events generated from screening | Over 3 years to determine long term outcomes from screening
  Adverse events generated from screening including incidental findings.
Assessment of the British Thoracic Society pulmonary nodule guidelines | Over 3 years to determine long term outcomes from screening
  Assessment of performance of the BTS pulmonary nodules guideline in the setting of screening service.
Smoking prevalence | Over 3 years to determine long term outcomes from screening
  Smoking prevalence and amount at the start and end of screening.
Undiagnosed airflow obstruction | Over 3 years to determine long term outcomes from screening
  Prevalence of undiagnosed airflow obstruction in the screened population.
Coronary artery calcification | Over 3 years to determine long term outcomes from screening
  Prevalence of coronary artery calcification and QRISK2 score.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Crosbie, Principal Investigator — Manchester University NHS Trust
Locations (1):
- Manchester University NHS Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only fully anonymised data will be sent to collaborating researchers